CLINICAL TRIAL: NCT02717104
Title: A Prospective, Multicenter, Single Arm, Post-Market Registry Assessing the Clinical Use and Safety of the LUTONIX Drug Coated Balloon Catheter in Femoropopliteal Arteries
Brief Title: Korean Post-market Registry Assessing the Clinical Use and Safety of the Lutonix DCB in Femoropopliteal Arteries
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: KORL15100
Record Dates: First submitted 2016-03-16; First posted 2016-03-23 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Artery Disease
Keywords: femoropopliteal
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the registry is to assess the clinical use and safety of the LUTONIX Drug Coated Balloon Catheter in a heterogeneous patient population in real world clinical practice.

DETAILED DESCRIPTION:
The registry will enroll patients with claudication or critical limb ischemia due to stenotic lesions in femoropopliteal arteries. All subjects meeting protocol criteria will be treated with the LUTONIX Drug Coated Balloon Catheter for approved indications according to the current Instructions for Use (IFU) and followed clinically for 2 years.

Total enrollment will be approximately 250 subjects at up to 18 sites. Subject follow-up will occur at 1, 6, 12 and 24 months. The primary efficacy endpoint is freedom from target lesion revascularization at 12 months.

The primary safety endpoint is freedom at 30 days from the composite endpoint of target vessel revascularization and target lesion revascularization, major amputation and major reintervention of index limb, and device- and procedure-related death.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years of age
* Rutherford Clinical Category ≥4
* Patient or Legally Authorized Representative is willing to provide informed consent and comply with the required follow-up
* Stenotic or obstructive vascular lesions in femoropopliteal artery(s)
* Lesion(s) can be treated with available LUTONIX Drug Coated Balloon Catheter device size matrix per current IFU
* At least one patent native outflow artery to the ankle free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of outflow disease is NOT permitted; treatment of in-flow disease is permitted prior to treatment with the LUTONIX Drug Coated PTA Dilatation Catheter)

Exclusion Criteria:

* Patient is currently participating in an active phase of another investigational drug or device study
* Inability to take recommended medications as stated in the IFU or non-controllable allergy to contrast
* Known inadequate distal outflow or planned future (within 30 days) treatment of vascular disease distal to the target lesion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General patient pool of participating hospitals or clinics
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Freedom from Target Lesion Revascularization | 12 months
Freedom from Target Vessel and Target Lesion Revascularization | 30 days
Freedom from Major Amputation and Major Reintervention of index limb | 30 days
Freedom from device- and procedure-related death | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kyu Kim, MD, Principal Investigator — Chonnam National University
Locations (16):
- South Korea (16):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Soonchunjyang University Hospital, Bucheon-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul, Jongno-gu
  - Busan Veterans Hospital, Busan
  - Inje University Busan Park Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - YeungNam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Konkuk University Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No